CLINICAL TRIAL: NCT04199858
Title: Electrophysiological Correlates of Nocebo Effects on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Universiteit Leiden (Other); VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, AWMEvers, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CEP19-1031/532
Record Dates: First submitted 2019-12-09; First posted 2019-12-16 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain Syndrome; Chronic Pain, Psychogenic; Chronic Pain; Hyperalgesia
Keywords: Pain; Nocebo; Hyperalgesia; Electroencephalography; EEG; Conditioning; Learning; Negative suggestions
MeSH Terms: conditions — Chronic Pain; Hyperalgesia; Pain

STUDY DESIGN:
Masking Description: A double-blind randomization list was created by an independent researcher to randomize participants into two counterbalanced conditions: participants either receive the nocebo sham medical gel in a blue or in a brown jar. Complete blinding of the researchers during the experiment is not possible due to the nature of conditioning/ suggestion paradigms. Participants are blind with respect to the conditioning/nocebo manipulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nocebo induction (Experimental): Conditioning and evocation of a nocebo response to a sham (inert) medication contained in a blue or a brown jar, controlled within subjects.
  Interventions: Behavioral: Baseline pain stimulations; Behavioral: Conditioning; Behavioral: Evocation; Other: Electroencephalography (EEG)

INTERVENTIONS:
Behavioral: Baseline pain stimulations — During baseline pain stimulations, a comparison block will include 6 high- and 2 moderate-pain stimulations.
Behavioral: Conditioning — During nocebo induction trials, the conditioned stimulus (i.e., a sham medical gel that can increase pain sensitivity, named "TDA" and contained in either a brown or a blue jar) is paired to unconditioned high-pain stimuli (nocebo trials). Lower 'baseline' pain is paired with no gel application (control trials).
  Other Names: Nocebo Induction phase
Behavioral: Evocation — During nocebo evocation, lower pain stimulations are administered both after the administration of the conditioned stimulus (i.e., a sham medical gel "TDA") and the control stimulus (no medical gel), in order to evoke nocebo responses to the sham hyperalgesic medication.
  Other Names: Nocebo testing phase
Other: Electroencephalography (EEG) — In the single group of participants, EEG recordings will be conducted during baseline, during a first resting-state of 5-minutes, during induction/evocation of nocebo responses, and during a second resting-state of 5-minutes.

SUMMARY:
Pain is a nociceptive somatosensory process that can arise as a debilitating and chronic symptom in various diseases or following an injury. How pain is experienced can vary widely within and across individuals, and can be shaped by cognitive processes such as learning. Nocebo effects, negative changes in symptom severity attributed to learned outcome-expectations, demonstrate how learning processes can be detrimental for the experience of pain. Research to date has produced inconclusive findings regarding the electrophysiological correlates on nocebo effects. The few studies that have applied electroencephalography (EEG) in this field have pointed towards a potential involvement of alpha-band activity, but the direction of this involvement remains unclear. For example, an EEG study of conditioned nocebo hyperalgesia found a pre to post increase in resting state alpha band power that was correlated with pain catastrophizing scores and not with the magnitude of the nocebo effect. Later, other studies also found pre to post changes in alpha band power, however, these changes were correlated with the magnitude of nocebo effects and not pain catastrophizing. Given the discrepancy in findings, in this study the investigators plan to primarily investigate whether EEG components predict the magnitude of nocebo responses to thermal-pain stimuli. The investigators will also explore electrophysiological correlates during pain anticipation and whether nocebo responses would be significantly related to spectral and temporal EEG biomarkers. This study will utilize a validated model of instructional and associative learning methods (i.e., negative suggestions and classical conditioning, respectively) to experimentally induce nocebo effects on heat-evoked pain. Developing objective, brain-derived markers for nocebo responses, or the detection of individuals most susceptible to nocebo hyperalgesia, will aid in the comprehensive management of pain. This study is conducted at Leiden University.

DETAILED DESCRIPTION:
Main outcome variable for nocebo responses:

- The magnitude of induced nocebo hyperalgesia is defined as the difference in pain ratings for the first nocebo trial compared to the first control trial of the evocation phase.

Note: A significant difference will be assessed using a Repeated Measures ANOVA as a manipulation check. Then, calculated difference scores represent the magnitude of induced nocebo hyperalgesia and will be used for the primary and first and second secondary hypotheses.

Definitions of other outcome variables:

- The magnitude of nocebo responses (and nocebo-augmented pain) during the evocation phase is defined in the specific nocebo evocation trials that show heightened pain relative to the preceding control trials, for each subject. For EEG analyses, all trials that show the experience of heightened pain in nocebo trials relative to the preceding control trials, during the evocation phase will be used.

Note: Calculated difference scores between the specific nocebo evocation trials that show heightened pain relative to control trials will be used in further analyses of EEG data. While the entirety of the evocation data will be reported and analyzed, the main EEG analyses will include a selection of evocation trials where nocebo responses were reported. It is necessary to use EEG data for trials that show a nocebo response in order to explore electrophysiological correlates of nocebo effects.

0. Manipulation checks: Induction of nocebo hyperalgesia First, the investigators will examine whether significant nocebo hyperalgesia was induced. A Repeated-Measures Analysis of Variance (RM ANOVA) will be performed for nocebo responses (on the pain Numeric Rating Scale), with trial type as the within-subjects factor with two levels (first nocebo evocation trial, first control evocation trial). First evocation trial pairs were chosen based on the clearest effects being observed during piloting and in previous nocebo studies.

1. Primary hypothesis:

   Pre-induction to post-induction decreases in resting-state alpha band power will positively correlate with the magnitude of induced nocebo hyperalgesia.
2. Secondary hypotheses:

   2.1. The magnitude of induced nocebo hyperalgesia in all nocebo-response evocation trials, will be related to temporal (e.g., Detrended Fluctuation Analysis) and spectral (e.g., Absolute Power, Relative Power and Central Frequency) biomarker values of alpha, beta, and gamma oscillations.

   2.2. The experience of nocebo-augmented pain in nocebo trials and pain during control trials of the evocation phase will be characterized by divergent alpha, beta, and gamma oscillation power and peak frequencies.

   2.3. The experience of nocebo-augmented pain in nocebo evocation trials and baseline high-pain stimulations, will be characterized by divergent alpha oscillation power and peak frequencies.

   2.4. The experience of control and nocebo trials during the induction phase, will be characterized by divergent alpha, beta, and gamma oscillation power and peak frequencies.

   2.5. Nocebo induction trials will be characterized by increased gamma band coherence relative to control induction trials during anticipation.
3. Questionnaires To assess the influence of psychological and personality traits, questionnaires will also be included. These will include the Pain Catastrophizing Scale (PSC), the Fear of Pain Questionnaire-III (FPQ-III), the Experience of Cognitive Intrusion of Pain (ECIP) scale, and the Amsterdam Resting State Questionnaire (ARSQ 2.0).

3.1. Correlation analyses will be performed between scores on the questionnaires and the magnitude of the nocebo effect.

3.2. Correlation analyses will be performed between scores on the questionnaires and measures of EEG, as well as pre-to post resting-state differences, in alpha, beta, and gamma frequency bands.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 35 years
* Good understanding of the English language
* Normal or corrected to normal vision

Exclusion Criteria:

* Ever having experienced serious medical or psychiatric conditions (e.g., heart or lung disease, panic attacks, drug addiction, clinical depression),
* Ever having experienced chronic pain complaints (pain for more than 6 months),
* Having experienced persisting painful health problems in the last 6 months,
* Experiencing acute physical pain (e.g., headache, or having used pain medication on the day of testing,
* Pregnancy or breastfeeding,
* Having recent injuries to the wrists or arms on the day of testing,
* Previous participation in this or similar studies (e.g., using conditioning or thermal pain).
* Having consumed psychotropic medication, recreational drugs, analgesic medication, or more than 3 units of alcohol, in the 24 hours prior to the study appointment.
* After inclusion, participants who do not reach a sensation of high pain (at least 6 on the NRS) with the highest administered temperature or participants will also be excluded.
* After inclusion, participants who do not reliably report a difference (a mean of at least 1,5 on the NRS) between the administered temperatures for control and nocebo trials in the induction phase will also be excluded. Nocebo conditioning relies upon the pairing of high-pain stimuli to the nocebo stimulus and lower pain to the control stimulus, therefore it is deemed that participants who do not experience this difference do not receive the necessary conditioning manipulation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants whose lived gender is male, will be included as male. Participants whose lived gender is female, will be included as female.
Enrollment: 36 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Magnitude of induced nocebo hyperalgesia | Through study completion, an average of 3 months
  The magnitude of induced nocebo hyperalgesia is defined as the difference in pain ratings for the first nocebo trial compared to the first control trial of the nocebo block evocation phase.
  A significant difference here is assessed within the mixed model ANOVA. Then, calculated difference scores represent the magnitude of induced effects and will be used in further analyses of EEG data.

SECONDARY OUTCOMES:
Magnitude of nocebo responses during evocation | Through study completion, an average of 3 months
  The magnitude of nocebo responses during the evocation phase is defined in the specific nocebo evocation trials that show heightened pain relative to control trials, for each subject.
Nocebo-augmented pain | Through study completion, an average of 3 months
  Nocebo-augmented pain is defined as the experience of heightened pain in nocebo trials relative to control trials, during the evocation phase.

OTHER OUTCOMES:
Electroencephalography components (EEG power in alpha band) | Through study completion, an average of 3 months
  Please refer to section Study Description / Detailed description.
Electroencephalography components (EEG power in beta band) | Through study completion, an average of 3 months
  Please refer to section Study Description / Detailed description.
Electroencephalography components (EEG power in gamma band) | Through study completion, an average of 3 months
  Please refer to section Study Description / Detailed description.
Electroencephalography components (EEG coherence in gamma band) | Through study completion, an average of 3 months
  Please refer to section Study Description / Detailed description.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea WM Evers, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data are collected pseudonymised thus no personal data are stored or shared. Consent forms are the only sources containing personal data and will not be shared, but are monitored by the department's Data Monitor.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available immediately after publication of the study and will be retained for 15 years.
Access Criteria: Data can be shared with scientists in relevant fields for the purpose of future studies such as replication or meta-analysis (or with designated persons for monitoring purposes).